CLINICAL TRIAL: NCT04931394
Title: A Prospective, Randomized, Controlled Trial of Adjuvant Chemotherapy for Pancreatic Cancer Based on Organoid Drug Sensitivity Test
Brief Title: Organoid-Guided Adjuvant Chemotherapy for Pancreatic Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Guo ShiWei, Associated Professor at the Institute of Pancreatic Surgery, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChanghaiH-PP08
Record Dates: First submitted 2021-06-15; First posted 2021-06-18 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Organoid; Drug Sensitivity Test; Chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Organoid-Guided Adjuvant Chemotherapy (Experimental): The pancreatic cancer specimens are obtained from surgery to be cultured for organoids. Then drug sensitivity is tested using organoid to obtain the sensitivity to the first-line drugs for pancreatic cancer (Gemcitabine, 5-fluorouracil, Paclitaxel, Oxaliplatin, Irinotecan). Patients will receive relatively sensitive chemotherapy regimen based on the test results. Adjuvant chemotherapy should start within 2 months after surgery, and last at least 6 months.
  Interventions: Other: Adjuvant chemotherapy guided by organoid drug sensitivity test
- Physician-decided Adjuvant Chemotherapy (No Intervention): The pancreatic cancer specimens are obtained from surgery to be cultured for organoids. Then drug sensitivity is tested using organoid to obtain the sensitivity to the first-line drugs for pancreatic cancer (Gemcitabine, 5-fluorouracil, Paclitaxel, Oxaliplatin, Irinotecan). Physician will decide the the adjuvant chemotherapy regimen, according to National Comprehensive Cancer Network (NCCN) guideline for pancreatic ductal adenocarcinoma. And they don't know the drug sensitivity test results. Adjuvant chemotherapy should start within 2 months after surgery, and last at least 6 months.

INTERVENTIONS:
Other: Adjuvant chemotherapy guided by organoid drug sensitivity test — Adjuvant chemotherapy guided by organoid will be given to pancreatic cancer patients.
  Arms: Organoid-Guided Adjuvant Chemotherapy

SUMMARY:
The purpose of this study is to explore whether adjuvant chemotherapy regimens guided by organoid drug sensitivity test can improve the outcomes of pancreatic cancer. At the same time, this study will evaluate the successful establishment rate of organoid from fresh surgical specimens , and explore the concordance between drug sensitivity test results and patients' treatment response.

DETAILED DESCRIPTION:
The poor prognosis of pancreatic cancer is not just because of the high malignancy of the tumor itself, but also its poor response to chemotherapy. At present, patient's drug-sensitivity is assessed by progression time after treatment. Therefore, it is difficult to judge a patient's sensitivity to a drug before adjuvant chemotherapy. Organoid is a new tumor model, which has the potential to test the drug sensitivity before chemotherapy.

Our center's previous experience has shown that the success rate of pancreatic cancer organoid culture is 77.6%. The previous research has confirmed that pancreatic cancer organoid was highly consistent with the original tissue in terms of genomics and histomorphology. More importantly, the investigators have tested the five first-line drug-sensitivity in 39 pancreatic cancer organoids, and compared the test results with the clinical treatment response of these patients, confirming that organoid can accurately evaluate the chemotherapy drug-sensitivity.

This is a single-center, prospective, open-label, randomized, controlled clinical trial, designed to explore whether adjuvant chemotherapy regimens guided by organoid drug sensitivity test can improve outcomes in pancreatic cancer patients. At the same time, the consistency between the drug sensitivity test results and the treatment response of patients will be analyzed. Also, the radiosensitivity of organoid will be tested, and be compared with the patients' response to radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years old and ≤80 years old.
* Complete R0 resection for pancreatic cancer with no evidence of malignant ascites, peritoneal metastases or distant metastases.
* Histology confirmed pancreatic adenocarcinoma.
* Eligible histologic variants include adenocarcinoma or variants to include mucinous adenocarcinoma or adenosquamous carcinoma.
* No metastases are found in preoperative examination.
* No prior chemotherapy or radiotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy of greater than 90 days, as judged by the investigator.
* Routine blood test: absolute neutrophil count>1500/mm3, platelet>100000/mm3.
* Normal liver function: serum total bilirubin≤2.0mg/dl, aminotransferase (ALT) and aspertate aminotransferase (AST) <2.5 times of the upper limit of normal value.
* Normal kidney function: serum creatinine<1.5 times of the upper limit of normal value or creatinine clearance rate>45ml/min.
* The pancreatic cancer organoid were cultured successfully.
* No severe comorbidities.

Exclusion Criteria:

* Patients with poor condition can not tolerate chemotherapy and targeted therapy.
* Impaired organ functions: heart failure (New York Heart Association III-IV), coronary heart disease, myocardial infarction within 6 months, severe cardiac arrhythmia and respiratory failure.
* Patients diagnosed with other cancer within 5 years.
* Patients who are pregnant or breastfeeding.
* Patients enrolled in other clinical trials or incompliant of regular follow up.
* Patients who did not provide an informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Disease free time | 1-2 years
  Time from the date of randomization to recurrence based on the radiology assessment of response using RECIST v1.1, or death, whichever is earlier.

SECONDARY OUTCOMES:
Overall survival time | 2-4 years
  The time from the date of randomization to the date of death for any cause. Patients will be followed until their date of death or until final database closure. Patients who are lost-to-follow-up or are alive at the time of analysis will be censored at the time they were last known to be alive or at the date of event cut-off for Overall survival (OS) analysis.
1-year disease-free survival | 1 year
  The percentage of patients without recurrence by one year.
The successful establishment rate of organoids | 2-4 years
  The rate of organoid successfully cultured in all the samples collected.
Concordance between drug sensitivity test results and patients' treatment response (descriptive statistics). | 2-4 years
  To assess the accuracy of drug sensitivity test in both group.The number of patients with correct prediction of treatment response by organoid drug-sensitivity test divided by the number of patients underwent chemotherapy.
Concordance between radiosensitivity test results and patients' treatment response (descriptive statistics). | 2-4 years
  To assess the accuracy of radiosensitivity test in both group. The number of patients with correct prediction of treatment response by organoid radiosensitivity test divided by the number of patients underwent radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Jin, M.D., Principal Investigator — Changhai Hospital, Shanghai, China
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No